CLINICAL TRIAL: NCT00586053
Title: "CTC of the Unprepped Colon: Optimization & Validation"
Brief Title: Unprepped CT Colonography
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: C. Daniel Johnson, M.D., Mayo Clinic
Other Study IDs: 1221-00; CA75333-08
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Colorectal Neoplasms
Keywords: Colonic Polyps; Colon; Large Intestine; Cecum; Sigmoid; Rectum; Colonoscopy; Virtual Colonoscopy; CT Colonography; Computed Tomographic Colonography; Colonography
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 485 patients,who have an average risk (asymptomatic and without colon screening in the last 5 years) or those who have a high risk for colon cancer (strong family history of colon cancer or polyps and/or personal history of colon cancer or polyps).
- 2: 160 patients, with a known colorectal lesion at or greater than 1 cm.
- 3: 610 patients, who are of average risk for colon cancer (asymptomatic and no colon cancer screening in the last 5 years).

SUMMARY:
It is our objective to improve the performance of CTC in the prepared colon, and to validate CTC in the unprepared colon for the detection of colorectal neoplasia. The cost-effectiveness ratio of CTC in the unprepared colon will compare favorably with other colorectal screening test.

DETAILED DESCRIPTION:
To improve the diagnostic performance of CTC in the prepared colon using improved spatial resolution, advanced image displays, and computer-assisted diagnosis, and to optimize diagnostic performance of CTC in the unprepared colon for colorectal polyp detection using electronic stool subtraction and computer-aided diagnostic techniques. To estimate the sensitivity and specificity of CTC in the unprepared colon for clinically important colorectal neoplasms (large adenomas ≥ 1 cm) and to compare such estimates with colonoscopy. To survey patient acceptance of CTC in the unprepared colon, and to assess implications for health care costs and cost-effectiveness of CTC in the unprepared colon in comparison with other approaches.

ELIGIBILITY:
Inclusion Criteria:

Average risk or higher for colorectal cancer and scheduled for colonoscopy with any of the following indications:

* Prior colorectal cancer, prior colorectal adenoma, strong family history of colorectal neoplasia, iron deficiency.
* Age ≥ 40 -100 years
* Known or highly suspected primary colorectal neoplasms > 10 mm (n = 160)
* Higher than average risk for colorectal cancer and scheduled for colonoscopy with any of the following indications: prior colorectal cancer, prior colorectal adenoma, strong family history of colorectal neoplasia, iron deficiency.

Exclusion Criteria:

* Less than 1/2 of colorectum remaining
* Inflammatory bowel disease (Crohns, Chronic Ulcerative Colitis)
* Familial Polyposis
* Melena, hematochezia

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic patients scheduled for colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 1255 (Actual)
Dates: Start 2000-08; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To optimize diagnostic performance of CTC in the unprepared colon for colorectal polyp detection using electronic stool subtraction and computer-aided diagnostic techniques. | 2000-2009

SECONDARY OUTCOMES:
The cost-effectiveness ratio of CTC in the unprepared colon will compare favorably with other colorectal screening tests | 2000-2009

CONTACTS AND LOCATIONS:
Overall Officials: C. Daniel Johnson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] MacCarty RL, Johnson CD, Fletcher JG, Wilson LA. Occult colorectal polyps on CT colonography: implications for surveillance. AJR Am J Roentgenol. 2006 May;186(5):1380-3. doi: 10.2214/AJR.05.0031. PMID 16632734
- [Result] Johnson CD, Fletcher JG, MacCarty RL, Mandrekar JN, Harmsen WS, Limburg PJ, Wilson LA. Effect of slice thickness and primary 2D versus 3D virtual dissection on colorectal lesion detection at CT colonography in 452 asymptomatic adults. AJR Am J Roentgenol. 2007 Sep;189(3):672-80. doi: 10.2214/AJR.07.2354. PMID 17715116